CLINICAL TRIAL: NCT05252416
Title: A Phase 1/2 Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of BLU-222 as a Single Agent and in Combination Therapy for Patients With Advanced Solid Tumors
Brief Title: (VELA) Study of BLU-222 in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This trial was terminated prior to the initiation of Phase 2 for reasons not due to safety concerns.
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BLU-222-1101
Record Dates: First submitted 2022-01-25; First posted 2022-02-23 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors; HR+ Breast Cancer; CCNE1 Amplification; HER2-negative Breast Cancer; Ovarian Cancer; Endometrial Cancer; Gastric Cancer; Esophageal Adenocarcinoma; Carcinosarcoma
Keywords: CDK2; CCNE1; Platinum-resistance; Platinum-refractory; CDK4/6i; Ribociclib; Carboplatin; Fulvestrant; ER+ Breast Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus; Carcinosarcoma | interventions — Carboplatin; ribociclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BLU-222 Monotherapy (Experimental): Dose Escalation: Multiple doses for BLU-222 for oral administration Dose Expansion: Oral dose of BLU-222 as determined during Dose Escalation
  Interventions: Drug: BLU-222
- BLU-222 + Carboplatin (Experimental): Dose Escalation: Multiple doses for BLU-222 for oral administration at doses deemed appropriate based on BLU-222 Monotherapy arm and multiple doses of Carboplatin at the approved dose.
  Dose Expansion: Oral dose of BLU-222 as determined during Dose Escalation and Carboplatin IV infusion at approved dose
  Interventions: Drug: BLU-222; Drug: Carboplatin
- BLU-222 + Ribociclib + Fulvestrant (Experimental): Dose Escalation: Multiple doses for BLU-222 for oral administration at doses deemed appropriate based on BLU-222 Monotherapy arm along with Ribociclib and Fulvestrant at the approved doses.
  Dose Expansion: Oral dose of BLU-222 as determined during dose escalation and approved doses of Ribociclib and Fulvestrant
  Interventions: Drug: BLU-222; Drug: Ribociclib; Drug: Fulvestrant
- BLU-222 + Fulvestrant (Experimental): Dose Expansion: Oral dose of BLU-222 as determined during Dose Escalation + fulvestrant at the approved dose
  Interventions: Drug: BLU-222; Drug: Fulvestrant

INTERVENTIONS:
Drug: BLU-222 — Oral administration
Drug: Carboplatin — IV Infusion
  Arms: BLU-222 + Carboplatin
Drug: Ribociclib — Oral administration
  Arms: BLU-222 + Ribociclib + Fulvestrant
Drug: Fulvestrant — Intra muscular administration
  Arms: BLU-222 + Fulvestrant; BLU-222 + Ribociclib + Fulvestrant

SUMMARY:
This is a Phase 1/2, open-label, first-in-human (FIH) study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and anticancer activity of BLU-222, a selective inhibitor of CDK2.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced solid tumors that has progressed beyond standard of care OR
2. HR+ HER2- BC that has progressed following treatment with a CDK4/6 inhibitor OR
3. Endometrial and gastric cancer that has progressed after at least 2 prior therapies (including one prior platinum therapy) OR
4. Platinum refractory or platinum resistant ovarian cancer CCNE1 amplified tumors that have progressed beyond standard of care

Exclusion Criteria:

1. Have visceral crisis, lymphangitic spread, or leptomeningeal carcinomatosis.
2. Have received the following anticancer therapy:

   a. Previous therapy with CDK2i, PKMYT1i, or WEE1i, except in Part 1A where up to 10 patients who previously received PKMYT1i, or WEE1 inhibitor will be permitted.
3. Have central nervous system (CNS) metastases or spinal cord compression that is associated with progressive neurological symptoms or requires increasing doses of corticosteroids to control the CNS disease.
4. Have known intracranial hemorrhage and/or bleeding diatheses.
5. Have clinically active ongoing ILD of any etiology, including drug-induced ILD, and radiation pneumonitis within 28 days prior to initiation of study treatment.
6. Have any unresolved toxicities from prior therapy greater than CTCAE Grade 1 or that have not resolved to baseline at the time of starting the study.
7. Have mean resting QTcF > 450 msec in men or QTcF > 470 msec in women, a history of prolonged QT syndrome or Torsades de pointes, or a familial history of prolonged QT syndrome.
8. Have clinically significant, uncontrolled, cardiovascular disease including congestive heart failure Grade III or IV according to the New York Heart Association classification; myocardial infarction or unstable angina within the previous 6 months, uncontrolled hypertension, or clinically significant, uncontrolled arrhythmias, including bradyarrhythmia that may cause QT prolongation (eg, Type II second degree heart block or third-degree heart block).
9. Have a history of another primary malignancy other than completely resected carcinomas in situ) that has been diagnosed or required therapy within 2 years prior to initiation of study treatment.
10. Have known active, uncontrolled infection (viral, bacterial, or fungal), including tuberculosis, hepatitis B virus (HBV), hepatitis C virus, AIDS-related illness, or COVID-19 infection (symptoms and a positive test result).
11. Requires treatment with a prohibited medication or herbal remedy that cannot be discontinued at least 2 weeks before the start of study drug administration.
12. Have planned major surgical procedure within 14 days of the first dose of study drug (procedures such as central venous catheter placement, tumor needle biopsy, and feeding tube placement are not considered major surgical procedures).
13. Unwilling or unable to comply with scheduled visits, study drug administration plan, laboratory tests, or other study procedures and study restrictions.
14. Patient is a woman who is not postmenopausal or surgically sterile, and is unwilling to abstain from sexual intercourse or employ highly effective contraception OR is a man who is not surgically sterile, and is unwilling to abstain from sexual intercourse or employ highly effective contraception
15. Patient is a pregnant female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
[Phase 1] Determine the maximum tolerated dose (MTD) of BLU-222 | Approximately 21 months
[Phase 1] Determine the recommended Phase 2 dose (RP2D) of BLU-222 | Approximately 21 months
[Phase 1] Rate and severity of adverse events | Approximately 21 months
[Phase 2] Overall response rate (ORR) | Approximately 43 months
[Phase 2] Rate and severity of adverse events | Approximately 43 months

SECONDARY OUTCOMES:
[Phase 1] Overall response rate (ORR) | Approximately 21 months
[Phase 1] Time of last quantifiable plasma drug concentration (Tlast) | Approximately 21 months
[Phase 1] Area under the plasma concentration time curve from time 0 to 12 hours (AUC0-12) | Approximately 21 months
[Phase 1] Area under the plasma concentration time curve from time 0 to 24 hours (AUC0-24) | Approximately 21 months
[Phase 1] Trough concentration (Ctrough) | Approximately 21 months
[Phase 1] Apparent volume of distribution (Vz/F) | Approximately 21 months
[Phase 1] Terminal elimination half-life (t½) | Approximately 21 months
[Phase 1] Apparent oral clearance(CL/F) | Approximately 21 months
[Phase 1] Accumulation ratio (R) | Approximately 21 months
[Phase 1] To assess treatment-induced modulation of biomarkers | Approximately 21 months
[Phase 1 and Phase 2] Duration of Response (DOR) | Approximately 43 months
[Phase 1 and Phase 2] Disease control rate (DCR) | Approximately 43 months
[Phase 1 and Phase 2] Clinical benefit rate (CBR) | Approximately 43 months
[Phase 1 and Phase 2] Progression free survival (PFS) | Approximately 43 months
[Phase 1 and Phase 2] Change in CA-125 levels | Approximately 43 months
[Phase 1 and Phase 2] Maximum plasma drug concentration (Cmax) | Approximately 43 months
[Phase 1 and Phase 2] Time to maximum plasma drug concentration (Tmax) | Approximately 43 months
[Phase 1 and Phase 2] Last measurable concentration (Clast) | Approximately 43 months
[Phase 1 and Phase 2] Area under the concentration-time curve from time 0 to the time of the last measured concentration AUC(0-last) | Approximately 43 months
[Phase 2] Overall survival (OS) | Approximately 43 months

CONTACTS AND LOCATIONS:
Locations (23):
- United States (19):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Women's Cancer Center, Stanford, California
  - Florida Cancer Specialists, Sarasota, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center (SKCCC), Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - UNC Hospitals at Chapel Hill - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Hospital of the Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah - Huntsman Cancer Institute - PPDS, Salt Lake City, Utah
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Instituto Europeo di Oncologia, Milan
  - Fondazione Policlinico Universitario A Gemelli-Rome, Rome
- St Bartholomew's Hospital, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No